CLINICAL TRIAL: NCT05291208
Title: Evaluation of a Cognitive Training Therapy Based on Synchronized Oscillatory Stimulation in Patients With Mild Cognitive Impairment Through a Randomized Clinical Trial
Brief Title: Clinical Trial Through Combined tACS Therapy in Patients With Mild Cognitive Impairment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad del Desarrollo (Other)
Responsible Party: Principal Investigator, Pablo Billeke, Social Neuroscience and Neuromodulation Laboratory Director, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SA19I0118
Record Dates: First submitted 2022-02-28; First posted 2022-03-22 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Mild Cognitive Impairment
Keywords: cognitive training; cognitive functions; non-invasive brain stimulation.; working memory
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): This group will receive a cognitive training intervention combined with alternating current electrical stimulation (i.e., treatment).
  Interventions: Combination Product: Combined tACS and Cognitive Training Program
- Control group (Sham Comparator): This group will receive a traditional cognitive training intervention with sham electrical stimulation.
  Interventions: Behavioral: Traditional Cognitive Training Program

INTERVENTIONS:
Combination Product: Combined tACS and Cognitive Training Program — The program contemplates 12 WM training sessions based on tasks of storage and manipulation of verbal and visuospatial information, with a frequency of twice a week during six weeks (total of 12 sessions). Patients will receive real electrical stimulation for 10 minutes during verbal working memory task. This includes 10s periods of phase-in and 10 s of phase-out and will be done in parallel with the cognitive intervention program in sessions 3, 4, 5, 6, 7, 8, 9, and 11. The electrical stimulation will be applied with two 3x1 arrays of electrodes. The central stimulation electrodes will be positioned in F3 and CP3 (10-20 system). The AC stimulation will be one mA from the baseline to the stimulation peak. The stimulation will have a gamma sine waveform (80Hz) over the positive phase of the theta oscillation (between 4 and 8 Hz, adjusted by each subject, Reinhart et al, 2019) phase-locked between arrays with impedances always under 10 kOhm.
  Arms: Treatment group
Behavioral: Traditional Cognitive Training Program — Participants will start a cognitive intervention program identical to the intervention group. Still, unlike the intervention group, they will receive placebo electrical stimulation, i.e., an electrical current will be applied for a short period at the beginning of the session (30 seconds), and then the stimulation will be stopped. This procedure induces a sensation in the skin similar to the real stimulation without generating a detectable impact on the brain state. They will be performed in parallel to the cognitive intervention program in sessions 1, 2, 3, 4, 5, 7, 9, and 10.
  Arms: Control group

SUMMARY:
The aging of the population has led to an increase in the prevalence of disabling and high-cost diseases, such as dementia and Mild Cognitive Impairment (MCI). The latter can be considered a prodromal phase of some dementias and a critical stage for interventions to postpone the impairment of functionality and thus maintain a better quality of life. A cognitive function to intervene in working memory (WM) since it represents the fundamental component of executive functions and is the gateway to maintaining long-term memory. This project proposes an intervention to enhance WM in these users, combining cognitive training with non-invasive brain stimulation, specifically transcranial electrical stimulation of alternating current (tACS). This proposal arises from recent evidence showing that it is possible to increase the capacity of WM in users with MCI through cognitive training. Along with this, tACS has been proposed as a specific neuronal plasticity inducer for the oscillatory pattern required for each mental process. WM is a process particularly susceptible to being enhanced by this technique, as the underlying electrophysiological oscillatory patterns of this process are well described. Thus, tACS would act as a potentiator of the residual capacity of WM in patients with neurodegenerative diseases.

This study is a phase II randomized, double-blind clinical trial with a 3-month follow-up. The study will be of 62 participants diagnosed with MCI over 60 years from Valparaíso, Chile. Participants will receive intervention that will combine 12 cognitive training sessions with non-invasive brain stimulation, specifically tACS. Depending on the intervention group to which they will be assigned, in 8 of these sessions, participants will receive either tACS or sham stimulation. Sessions will last approximately 1 hour and take place twice a week, over six weeks. The primary outcomes will be the electroencephalographic measurements, and the secondary effects will be cognitive assessments of WM. The outcomes will be performed before, immediately after, and three months after the end of the intervention.

The outcomes of this trial will add evidence about the benefits and feasibility of an intervention that combines cognitive training with non-invasive brain stimulation. The objective is to contribute tools for optimal cognitive treatment in patients with MCI. To enhance WM capacity, postpone the impairment of functionality, and obtain a better quality of life.

DETAILED DESCRIPTION:
Background At the global level, sociodemographic change is happening, characterized by progressive aging of the population and a modification of the epidemiological profile, with an increase in the prevalence of chronic diseases and other pathologies associated with aging, such as dementia. Dementia is an acquired and chronic pathology characterized by an impairment of brain functions involving cognitive, psychological, and behavioral symptoms. These symptoms affect people's ability to carry out their usual daily activities. These disabilities imply a challenge for the people themselves, their families, the state, and public policies.

To date, the therapeutic approach to patients with dementia has focused primarily on late-stage drug treatment. However, this type of intervention has reported good results on specific dimensions, and an efficacy questioned long-term. The use of drugs with non-pharmacological therapies has proposed that it would be more effective to complement the treatment of patients, and the efforts should be directed towards prevention. In this context, in prodromal phases of dementia, such as Mild Cognitive Impairment (MCI), it is suggested early interventions.

MCI refers to the intermediate stage between the cognitive changes observed by normal aging and those that occur due to dementia. Patients with MCI are especially likely to benefit from non-pharmacological intervention. Since these patients would maintain some degree of neuroplasticity, the patients would learn and apply new strategies to improve their cognitive functioning.

One critical component of cognitive skills affected in neurodegenerative diseases and dementias is working memory (WM). WM represents a fundamental pillar of cognitive functions and is the gateway to the maintenance of long-term memory. The traditional view assumes that the capacity of WM is a specific feature of each individual and that it is not modifiable. However, recent evidence has accumulated that the capacity of WM is susceptible to be enhanced by training. This improvement is related to enhanced activity, connectivity, and selectivity between the frontal and parietal cortex.

Despite these findings, most evidence comes from healthy populations with conserved neuroplasticity. This constitutes a problem for neurodegenerative diseases because it has been corroborated that neuroplasticity is limited in these pathologies. In this context, cognitive rehabilitation in these diseases must include therapeutic tools aimed at increasing neuroplasticity. The use of non-invasive brain stimulation offers an opportunity to increase the capacity of neuroplasticity in this population. However, there has not been a rehabilitation proposal that incorporates this technique into intervention programs. Advancements have been made in neuroscience on the mechanisms underlying WM that have not been incorporated into early intervention and cognitive training in subjects with MCI.

Some studies have shown that it is possible, on the one hand, to preserve cognitive abilities in these patients, avoiding conversion to dementia and, on the other hand, the reversibility of a certain degree of impairment. Also, there is evidence of the influence of environmental and lifestyle factors as protective and moderating agents in maintaining cognitive skills. It seems logical to propose cognitive training as a preventive factor and as a therapeutic tool along these lines. In neurophysiological terms, it has been observed that patients with MCI exhibit disruptions in brain oscillations, which are similar to those observed in patients with dementia. And these altered brain oscillatory patterns are at the basis of cognitive alteration evidenced in this pathology.

Based on these disturbances oscillatory patterns, it is possible to propose non-invasive brain stimulation. Indeed, transcranial electrical stimulation (tES) is a safe tool widely used in research and validated for clinical use in both healthy subjects and patients. This technique modulates neuronal excitability without directly generating an action potential. Using this is called transcranial alternating current stimulation (tACS) in an oscillatory manner. This technique causes changes by increasing the specific oscillatory activity in the existing neuronal circuits that underlie a cognitive process. And, the enhancement in these oscillatory patterns triggers an increase in neuroplasticity. In this context, WM is a process that is particularly amenable to being enhanced with this technique, as the underlying electrophysiological patterns have been described.

Neuroimaging and brain electrical activity studies show that WM depends on distributed functional networks that involve an oscillatory activity in different ranges of frequency, mainly involving fronto-parietal association cortices.

The implementation of WM training improves its performance, and it has been associated with increased activity, connectivity, and selectivity, mainly of the frontal and parietal association cortices. As fronto-parietal networks are involved in diverse cognitive tasks, training could explain the transfer effect of WM training on improving functionality in daily life. To date, initiatives proposing interventions that add cognitive training and facilitate neuroplasticity in subjects with MCI are scarce. However, there is scientific and clinical interest in finding conclusive evidence in this regard, which is currently demonstrated by two registered clinical trials.

These studies reinforce the need to develop evidence concerning therapeutic alternatives that impact users' quality of life, thus reducing their degree of cognitive disability. In this context, it is proposed to evaluate the effect of a WM training therapy, which involves theta-band synchronic tACS on the prefrontal and parietal regions, in a group of users with MCI compared to an intervention involving only cognitive training.

Methods and design This study has a parallel design, where two groups will receive two different interventions. The investigator will study the characteristics of the factors and effects. In this manner, this analysis allows us to conceptualize the design as a 2x3 mixed factorial. Thus, The investigator will include a factor between groups (type of intervention, two levels) and an intra-subject factor (two dependent variable measurements will be implemented in three episodes, one pre-intervention and two post-intervention). This type of design will allow studying the potential interaction effects between the inter and intra-subject factors.

Participants The study's target population will be non-institutionalized users with Mild Cognitive Impairment referred to the Center of Phonoaudiological Attention of the University of Valparaiso from Valparaiso, Chile. The recruitment of participants will be done by a clinical team consisting of a neuropsychologist, a clinical psychologist, and speech therapists, who will apply the instruments to corroborate the fulfillment of the inclusion-exclusion criteria. In addition, the clinical team will carry out the evaluations and interventions that the participants will receive once these users have expressed their willingness to participate in the study by signing informed consent. For the estimation of the minimum required sample size, the investigators consider the following parameters: a) Effect size for the mixed ANOVA statistical test (2 x 2, with interaction effects), b) Statistical power (1- Beta)=.95 and c) Significance level alpha=.05. The investigators used the G*Power 3 software to calculate. Considering an effect size n2 =0.06, the sample size amounts to a total of 54 participants (n1=27; n2=27). As our study was a two intervention effect, the investigators considered an effect size somewhat smaller than those observed for comparisons between clinical populations of prefrontal theta oscillations during working memory: for example Lenartowicz, et al., 2014 : n2 =0.09, and which coincides with the work of our team, Larrain-Valenzuela 2017; Figuera et al., 2020 n2 ~ 0.1. The effect size that the investigators used to calculate the sample is considered a moderate to large effect according to Cohen's criteria (1988). This criterion is vital if the investigators consider the importance of finding effects that are only statistically significant but also clinically relevant. However, the initial sample size that the investigators propose in this project will consider the proportion of participants who may present low adherence to the study. In this regard, the investigators can point out that in a preliminary study (IUD-65/13) with similar characteristics, a drop-out rate of about 15% was observed. Therefore, considering the drop-out percentage and the minimum sample size required to investigate an effect, the initial sample will be 62 participants (n1=31; n2=31).

Procedure This clinical trial will randomize using the stratified randomization method, whose strata will be age (<75 years and >=75 years), sex (male and female) and educational levels (<=12 years of education and >12 years of educations). After stratification, simple randomization will be use. Each participant will have the same probability of being assigned to either of the two intervention groups. For this purpose, the table of random numbers will be used as a base tool through a computer system available. The person in charge of generating the random assignment sequence list will be unaware of the people who recruit and evaluate the participants.

Data analysis Inferential Analysis. Compliance with assumptions for parametric testing will be contrasted. In particular, univariate normality (i.e., Kolmogorov-Smirnoff, Shapiro-Wilk), sphericity (i.e., Mauchly's W), and homoscedasticity of error variances (i.e., Levene test). If any of the above assumptions are violated, the corresponding non-parametric estimates will be provided. Once the assumptions have been tested, the data analysis includes the mixed ANOVA test with interaction effects. The following parameters will be evaluated in the model: (a) main effects of the factor between groups, (b) main effects of the factor within groups, and (c) interaction effects between inter and intra factors. For each electrophysiological and cognitive performance measure analysis, the respective effect size will be reported through each analysis's index n2p (partial eta square). The respective post hoc comparisons will use Bonferroni's correction, and the respective effect size will be reported through Cohen's index d. Graphs of the interaction effects will be provided if observed. In case of transgression of the sphericity assumption, the Greenhouse-Geisser correction will be made. Consequently, the respective parametric statistics will be provided (i.e., Friedman test, Connover's Post hoc tests). For all hypothesis tests, a significance level will be considered alpha=.05.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 60 years.
* Presence of Mild Cognitive Impairment, according to the diagnostic criteria established in Petersen et al. (2014).
* Have six or more years of complete schooling (presence of reading and writing).

Exclusion Criteria:

* The previous diagnosis of other neurodegenerative diseases.
* Attending another cognitive training program.
* History of Epilepsy or current presence of epileptic seizures.
* Presence of psychiatric diseases.
* Presence of a relevant depressive picture (GDS >=2).
* History of important neurological alterations such as the history of stroke, transient ischemic attack, cranial brain trauma.

Important alterations of communication.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-09-21 (Estimated); Study Completion 2024-09-21 (Estimated)

PRIMARY OUTCOMES:
Prefrontal theta oscillation activity. | week 1 (pre-intervention), week 8 (1 week post intervention), week 20 (12 weeks post intervention)
  The ratio of change of the normalized power (mean/standard error, micro Volt2 ) of prefrontal theta oscillation (5-10 Hz, Fz electrode) related to Successful Memory Performance. The prefrontal theta oscillation related to Successful Memory Performance (SMP) is calculated based on a single-trial general linear model that include SMP as the regressor of interest and Memory Load as a secondary regressor.

SECONDARY OUTCOMES:
WAIS-IV Digit Retention subtest. Chilean standard. (Rosas et al., 2015) | week 1 (pre-intervention), week 8 (1 week post intervention), week 20 (12 weeks post intervention)
  It is part of the Working Memory Index and consists of three tasks: a) Direct Digits: repeat a series of digits, presented orally, in the same order as they are presented; b) Reverse Order Digits: repeat a series of digits in reverse order of presentation; and c) Sequence Digits: order and repeat from lowest to highest a series of numbers read by the examiner. These tasks assess attention and resistance to distraction, immediate auditory memory, and working memory (i.e., reverse order, sequence).
Trail Making Test B (TMT-B). Chilean standard. (Arango-Lasprilla et al., 2015) | week 1 (pre-intervention), week 8 (1 week post intervention), week 20 (12 weeks post intervention)
  TMT - B. This part of TMT reflects mainly working memory and secondarily the capacity for cognitive flexibility. It connects 25 numbers and letters in ascending order, alternating between them (e.g., 1-A, 2-B, 3-C, etc.). The score is obtained from the time it takes an individual to complete the task.
Parietal theta oscillation activity. | week 1 (pre-intervention), week 8 (1 week post intervention), week 20 (12 weeks post intervention)
  The ratio of change of the normalized power (mean/standard error, micro Volt2 ) of parietal theta oscillation (5-10 Hz, CP3 electrode) related to Memory Load. The parietal theta oscillation related to Memory Load is calculated based on a on a single-trial general linear model that include Memory Load as the regressor of interest and Successful Memory Performance (SMP) as a secondary regressor.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Billeke, PhD, Principal Investigator — Social Neuroscience and Neuromodulation Laboratory Director
Locations (1):
- Centro de Investigación del Desarrollo de Cognición y Lenguaje, Faculty of Medicine, Universidad de Valparaíso., Valparaíso, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alekseichuk I, Turi Z, Amador de Lara G, Antal A, Paulus W. Spatial Working Memory in Humans Depends on Theta and High Gamma Synchronization in the Prefrontal Cortex. Curr Biol. 2016 Jun 20;26(12):1513-1521. doi: 10.1016/j.cub.2016.04.035. Epub 2016 May 26. PMID 27238283
- [Background] Arango-Lasprilla JC, Rivera D, Aguayo A, Rodriguez W, Garza MT, Saracho CP, Rodriguez-Agudelo Y, Aliaga A, Weiler G, Luna M, Longoni M, Ocampo-Barba N, Galarza-Del-Angel J, Panyavin I, Guerra A, Esenarro L, Garcia de la Cadena P, Martinez C, Perrin PB. Trail Making Test: Normative data for the Latin American Spanish speaking adult population. NeuroRehabilitation. 2015;37(4):639-61. doi: 10.3233/NRE-151284. PMID 26639932
- [Background] Babiloni C, Del Percio C, Pascarelli MT, Lizio R, Noce G, Lopez S, Rizzo M, Ferri R, Soricelli A, Nobili F, Arnaldi D, Fama F, Orzi F, Buttinelli C, Giubilei F, Salvetti M, Cipollini V, Franciotti R, Onofrj M, Stirpe P, Fuhr P, Gschwandtner U, Ransmayr G, Aarsland D, Parnetti L, Farotti L, Marizzoni M, D'Antonio F, De Lena C, Guntekin B, Hanoglu L, Yener G, Emek-Savas DD, Triggiani AI, Taylor JP, McKeith I, Stocchi F, Vacca L, Hampel H, Frisoni GB, De Pandis MF, Bonanni L. Abnormalities of functional cortical source connectivity of resting-state electroencephalographic alpha rhythms are similar in patients with mild cognitive impairment due to Alzheimer's and Lewy body diseases. Neurobiol Aging. 2019 May;77:112-127. doi: 10.1016/j.neurobiolaging.2019.01.013. Epub 2019 Jan 24. PMID 30797169
- [Background] Constantinidis C, Klingberg T. The neuroscience of working memory capacity and training. Nat Rev Neurosci. 2016 Jul;17(7):438-49. doi: 10.1038/nrn.2016.43. Epub 2016 May 26. PMID 27225070
- [Background] George MS, Aston-Jones G. Noninvasive techniques for probing neurocircuitry and treating illness: vagus nerve stimulation (VNS), transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS). Neuropsychopharmacology. 2010 Jan;35(1):301-16. doi: 10.1038/npp.2009.87. PMID 19693003
- [Background] Larrain-Valenzuela J, Zamorano F, Soto-Icaza P, Carrasco X, Herrera C, Daiber F, Aboitiz F, Billeke P. Theta and Alpha Oscillation Impairments in Autistic Spectrum Disorder Reflect Working Memory Deficit. Sci Rep. 2017 Oct 30;7(1):14328. doi: 10.1038/s41598-017-14744-8. PMID 29085047
- [Background] Melloni M, Billeke P, Baez S, Hesse E, de la Fuente L, Forno G, Birba A, Garcia-Cordero I, Serrano C, Plastino A, Slachevsky A, Huepe D, Sigman M, Manes F, Garcia AM, Sedeno L, Ibanez A. Your perspective and my benefit: multiple lesion models of self-other integration strategies during social bargaining. Brain. 2016 Nov 1;139(11):3022-3040. doi: 10.1093/brain/aww231. PMID 27679483
- [Background] Soto-Icaza P, Vargas L, Aboitiz F, Billeke P. Beta oscillations precede joint attention and correlate with mentalization in typical development and autism. Cortex. 2019 Apr;113:210-228. doi: 10.1016/j.cortex.2018.12.018. Epub 2019 Jan 2. PMID 30677619
- [Background] Reinhart RMG, Nguyen JA. Working memory revived in older adults by synchronizing rhythmic brain circuits. Nat Neurosci. 2019 May;22(5):820-827. doi: 10.1038/s41593-019-0371-x. Epub 2019 Apr 8. PMID 30962628
- [Background] Figueroa-Vargas A, Carcamo C, Henriquez-Ch R, Zamorano F, Ciampi E, Uribe-San-Martin R, Vasquez M, Aboitiz F, Billeke P. Frontoparietal connectivity correlates with working memory performance in multiple sclerosis. Sci Rep. 2020 Jun 9;10(1):9310. doi: 10.1038/s41598-020-66279-0. PMID 32518271
- [Background] Billeke P, Armijo A, Castillo D, Lopez T, Zamorano F, Cosmelli D, Aboitiz F. Paradoxical Expectation: Oscillatory Brain Activity Reveals Social Interaction Impairment in Schizophrenia. Biol Psychiatry. 2015 Sep 15;78(6):421-31. doi: 10.1016/j.biopsych.2015.02.012. Epub 2015 Feb 19. PMID 25861703
- [Background] Martin DM, Liu R, Alonzo A, Green M, Player MJ, Sachdev P, Loo CK. Can transcranial direct current stimulation enhance outcomes from cognitive training? A randomized controlled trial in healthy participants. Int J Neuropsychopharmacol. 2013 Oct;16(9):1927-36. doi: 10.1017/S1461145713000539. Epub 2013 May 30. PMID 23719048
- [Derived] Figueroa-Vargas A, Gongora B, Alonso MF, Ortega A, Soto-Fernandez P, Z-Rivera L, Ramirez S, Gonzalez F, Munoz Venturelli P, Billeke P. The effect of a cognitive training therapy based on stimulation of brain oscillations in patients with mild cognitive impairment in a Chilean sample: study protocol for a phase IIb, 2 x 3 mixed factorial, double-blind randomised controlled trial. Trials. 2024 Feb 23;25(1):144. doi: 10.1186/s13063-024-07972-7. PMID 38395980